CLINICAL TRIAL: NCT07322783
Title: Osimertinib Combined With Savolitinib in the Treatment of EGFR Mutated Osimertinib Resistant NSCLC With Low Copy Number MET Amplification
Brief Title: Osimertinib Combined With Savolitinib in the Treatment of NSCLC With Low Copy Number MET Amplification
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Qingdao Central Hospital (Other)
Responsible Party: Principal Investigator, Youxin Ji, President, Qingdao Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY202512203
Record Dates: First submitted 2025-12-16; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: EGFR Positive Non-small Cell Lung Cancer; MET Amplification
Keywords: Savolitinib; Osimertinib; Drug Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Savolitinib plus osimertinib (Experimental)
  Interventions: Drug: • Drug: Savolitinib • Drug: Osimertinib Mesylate Tablets

INTERVENTIONS:
Drug: • Drug: Savolitinib • Drug: Osimertinib Mesylate Tablets — Osimertinib 80 mg oral daily, savolitinib 400-600 mg (400mg for body weight <60 kg, 600 mg for body weight >60 kg) until disease progression or intolerable toxicities. Dose reduction of savolitinib can be from 600 mg to 400 mg and 400 mg to 200 mg.

SUMMARY:
Osimertinib combined with savolitinib in the treatment of EGFR mutated osimertinib resistant NSCLC with low copy number MET amplification There are unmet medical needs in patients who resist to to osimertinib; savolitinib plus osimertinib shows high response rate and prolong progression-free survival in high copy number MET amplification patients. This study is to explore the efficacy and safety of the combination of savolitinib and osimertinib in osimertinb resistant patients with low copy number MET amplification.

DETAILED DESCRIPTION:
his is an open-label, single-arm, multicenter, phase 2 study. Low copy number MET amplification is defined as MET amplification copy number below 5 tested with NGS or FISH. All patients were 3rd or more lines therapy that had resistant to osimertinib, chemo-immunotherapy or anti-angiogenesis. Osimertinib mesylate tablets (hereinafter referred to as osimertinib) is 80 mg oral daily, savolitinib 400-600 mg (400mg for body weight <60 kg, 600 mg for body weight >60 kg) until disease progression or intolerable toxicities. Dose reduction of savolitinib can be from 600 mg to 400 mg and 400 mg to 200 mg.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically or cytologically confirmed incurable advanced or metastatic non-small cell lung cancer who resistant to resistant to osimertinib, chemo-immunotherapy or anti-angiogenesis.

  2. At least 1 measurable lesion (RECIST 1.1). 3. MET amplification copy number below 5 by FISH. 4. Male or female patients age ≥18 years. 5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2. 6. Estimated OS ≥3 months. 7. Adequate hematologic and bone marrow functions. 8. Adequate renal and liver function. 9. Had recovered from all toxicities related to prior anticancer therapies to grade ≤ 2, except for patients with grade 2 nausea/vomiting and/or grade 2 diarrhea despite optimal supportive therapy who will not be allowed to participate in the study.

  10. Willingness to use contraception by a method that is deemed effective by the investigator by both males and female patients of child bearing potential (postmenopausal women must have been amenorrhea for at least 12 months to be considered of non-childbearing potential) and their partners throughout the treatment period and for at least three months following the last dose of study drug.

  11. Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the patient prior to any study-specific procedures).

  12. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion13. Any of the following cardiac criteria: screening period resting period QTC > 470 milliseconds (clinical electrocardiograph report value; if a single time> 470 milliseconds, take the average of 3 inspections); rhythm of resting electrocardiogram (ECG), any clinically important abnormality of conduction or morphology (e.g., complete left bundle branch block, Grade 3 heart block, Grade 2 heart block); family history of congenital long QT prolongation syndrome or long QT syndrome.

14. Evidence of any serious or uncontrolled systemic disease; various chronic active infections such as hepatitis B (HBV-DNA ≥ 104 copy number/ml or 2000 IU/ml), hepatitis C and HIV; uncontrollable Hypertensive patients (requires 2 or more drugs to control blood pressure); unstable angina; angina pectoris within 3 months prior to study; congestive heart failure (NYHA class II or higher); myocardial infarction (NSTEMI or STEMI) history in 6 months before study enrollment; severe arrhythmia requiring medical attention; severe liver, kidney, gastrointestinal or metabolic diseases.

15. Patients who are unable to taking drugs 16. Other malignancies need treatment; except effectively treated skin basal cell carcinoma, cutaneous squamous cell carcinoma, and/or effectively resected orthotopic cervical cancer and/or breast cancer.

17. Female patients during pregnancy or lactation. 18. Previous allergies or intolerance to treatment with osimertinib and savolitinib.

19. Any other condition or circumstance of that would, in the opinion of the investigator, make the patient unsuitable for participation in the study.

Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | the percentage of patients getting partial response and complete response, assessed at 2 month.
  Overall response rate defined as the percentage of patients getting partial response and complete response after treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of enrollment until the date of disease progression of patient death from any cause, assessed up to 24 months
  Progression-free survival is defined as the time from the date of enrollment to the date of disease progression or patient death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Qingdao Central Hospital, Qingdao, China